CLINICAL TRIAL: NCT03926156
Title: RIvoraxaban Safety and Efficacy in Patients With Mitral Stenosis
Brief Title: RIvoraxaban in Mitral Stenosis
Acronym: RISE MS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID-19 has impacted our study recruitment
Sponsor: Rajaie Cardiovascular Medical and Research Center (Other)
Collaborators: National Institute for Medical research and Development (NIMAD) (Unknown); Abidi Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 962426
Record Dates: First submitted 2019-04-22; First posted 2019-04-24 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Mitral Stenosis; Rheumatic Heart Disease; Atrial Fibrillation; Anticoagulant Adverse Reaction
MeSH Terms: conditions — Mitral Valve Stenosis; Rheumatic Heart Disease; Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Experimental): Rivaroxaban will be used as the anticoagulation drug for the intervention group. Rivaroxaban is an anticoagulant and the first orally active direct factor Xa inhibitor. Unlike warfarin, routine lab monitoring of INR is not necessary. However there is no approved antidote available in the event of a major bleed. Only the 10 mg tablet can be taken without regard to food. The 15 mg and 20 mg tablet should be taken with food.
  Interventions: Drug: Rivaroxaban
- Warfarin (Active Comparator): Warfarin will be used as the anticoagulation drug for the control group. Warfarin decreases blood clotting by blocking an enzyme called vitamin K epoxide reductase that reactivates vitamin K1. Without sufficient active vitamin K1, clotting factors II, VII, IX, and X have decreased clotting ability. The anticlotting protein C and protein S are also inhibited but to a lesser degree. A few days are required for full effect to occur and these effects can last for up to five days, and the final dose will be adjusted according to PT and related INR.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban — Rivaroxaban will be used as the anticoagulation drug for the intervention group. Rivaroxaban is an anticoagulant and the first orally active direct factor Xa inhibitor. Unlike warfarin, routine lab monitoring of INR is not necessary. However there is no approved antidote available in the event of a major bleed. Only the 10 mg tablet can be taken without regard to food. The 15 mg and 20 mg tablet should be taken with food
  Arms: Rivaroxaban
Drug: Warfarin — Warfarin will be used as the anticoagulation drug for the control group. Warfarin decreases blood clotting by blocking an enzyme called vitamin K epoxide reductase that reactivates vitamin K1. Without sufficient active vitamin K1, clotting factors II, VII, IX, and X have decreased clotting ability. The anticlotting protein C and protein S are also inhibited but to a lesser degree. A few days are required for full effect to occur and these effects can last for up to five days, and the final dose will be adjusted according to PT and related INR.
  Arms: Warfarin

SUMMARY:
In this randomized controlled clinical trial, patients with moderate to severe mitral valve stenosis (MS) and atrial fibrillation (AF) will be enrolled into the study.Participants will be divided into two groups based on the anticoagulation regimen type. The intervention group will receive rivaroxaban and the control group will be given warfarin. All patients will be observed closely during a period of one year. Through the follow up, embolic events and hemorrhagic complications will be recorded in both groups. In addition, patients in both group will undergo a baseline magnetic resonance imaging (MRI) and an MRI after one-year follow up, by which the silent embolic events will be compared in both groups.

DETAILED DESCRIPTION:
Study rationale:

Since the introduction of warfarin as the main oral anticoagulation therapy in patients with MS and AF, no other drug has been replaced/suggested by any medical community for this group of patients. Warfarin is considered a drug with marginal therapeutic effect, with a need for constant monitoring, with lots of known drug interaction and finally a great probability of adverse complication. Novel oral anticoagulation agents have resolved several of these drawbacks and has been recommended as a viable option as a substitute of warfarin in various clinical scenario. Until now, no trial has evaluated the potentiality of using novel oral anticoagulations (NOACs) in patients with MS accompanied by AF. In this trial investigators are intended to elaborate the efficacy and safety of rivaroxaban in patients with MS complicated by AF

Background:

Since the introduction of NOAC, their indication has been expanded in various type of diseases. From protecting against ischemic stroke in AF patients to treatment of venous thromboembolism (VTE) events, NOAC were both safe and effective compared to warfarin. Importantly this new class of drug have omitted some of the major drawbacks of warfarin; their predictable therapeutic level has permitted to prescribed them as fixed dosage without constant laboratory tests. Also their shorter half-life has made critical situation in which reversal of anticoagulation agents were needed, more manageable.

There are solid evidences that AF is one of the major cause of cerebrovascular ischemic events, and anticoagulation therapy by decreasing thrombus formation reduces significantly these major adverse events. So there is no wonder that first studies on NOAC were performed on AF population. In the beginning AF caused by valvular heart diseases were judge to bear a much greater risk as cerebrovascular events are concerns, and consequently patients with valvular pathologies were eliminated from the earlier pivotal studies. However, through these years, there are lots of evidences showing the safety and efficacy of NOAC in valvular pathologies. Recently ENGAGE TIMI 48 Trial has showed the efficacy and safety of Edoxaban in patients with valvular heart diseases. By testing the theory in a large population, the ENGAGE TIMI 48 study emphasized on a greater risk of embolic events in patients with VHD and AF, but this increasing risk has no effect on the efficacy of edoxaban compared to warfarin. Interestingly the new agents had less major bleeding compared to warfarin.

But still in all these trials, moderate to severe MS and mechanical prosthetic valves were omitted from the studied population. The rationale behind this omission was the significant higher risk of thrombosis in the two mentioned subgroups. However, investigators have several hypotheses that patients with MS are different from patients undergoing mechanical prosthetic valve replacement:

* Although there is a higher risk of thromboembolic events in MS comparing to other valvular heart diseases, this has not resulted in increasing the magnitude of protection with warfarin; the recommended levels of international normalized ratio (INR) in MS population is 2-3 as other pathologies.
* Apart from patients with mechanical prosthesis implanted in mitral valve position, there is no other subgroup of patients whom higher INR and level of anticoagulation with warfarin proved to be more efficacious.

In conclusion, investigators think that the MS population might be a good target for NOAC and as other valvular heart disease, they could benefit from the advantages of these drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Men and women ≥ 18 year-old
4. Diagnosed with moderate to severe mitral stenosis who have a history of AF of any duration documented by any electrical tracing within the prior 12 months and for which anticoagulation is indicated and planned for the duration of the study.
5. Ability to take oral medication and be willing to adhere to the rivaroxaban regimen

Exclusion Criteria:

1. Left atrial clot
2. Severe renal dysfunction (creatinine clearance [CrCl] <15 mL/min), subjects with
3. A condition associated with a high risk of bleeding
4. Allergic to rivaroxabn/warfarin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with stroke | 12 months
  A stroke is defined as an abrupt onset, over minutes to hours, of a focal neurological deficit in the distribution of a single brain artery that is not due to an identifiable nonvascular cause (i.e., brain tumor or trauma), and that either lasts at least 24 hours or results in death within 24 hours of onset.
Number of participants with systemic embolic event | 12 months
  An SEE is defined as an arterial embolism resulting in clinical ischemia, excluding the central nervous system (CNS), coronary and pulmonary arterial circulation.

SECONDARY OUTCOMES:
Number of participants with bleeding complications | 12 months
  Bleeding complication will be assessed according to the International Society on Thrombosis and Haemostasis.

CONTACTS AND LOCATIONS:
Overall Officials: Majid Maleki, M.D., Study Chair — Rajaie Cardiovascular Medical and Research Center
Locations (1):
- Rajaie Cardiovascular Medical and Research Center, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sadeghipour P, Pouraliakbar H, Parsaee M, Shojaeifard M, Farrashi M, JamalKhani S, Tashakori Beheshti A, Rostambeigi S, Ebrahimi Meimand S, Firouzi A, Peighambari MM, Alemzadeh-Ansari MJ, Haghjoo M, Noohi F, Maleki M, De Caterina R. RIvaroxaban in mitral stenosis (RISE MS): A pilot randomized clinical trial. Int J Cardiol. 2022 Jun 1;356:83-86. doi: 10.1016/j.ijcard.2022.03.037. Epub 2022 Mar 16. PMID 35306032